CLINICAL TRIAL: NCT04905576
Title: Quality of Life Interventions During Cervical Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Susan Lutgendorf, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 200105058
Record Dates: First submitted 2021-05-20; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; healing touch; healing touch therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Relaxation Therapy; Therapeutic Touch; Touch; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Patients are randomized to relaxation, healing touch, or standard care arms of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Relaxation training following daily radiation (Experimental): All relaxation sessions will be given individually, and will be provided by trained nurses or research assistants. Patients receiving relaxation will learn exercises to release tension through muscle relaxation, breathing, and imagery
  Interventions: Behavioral: Relaxation training; Other: Questionnaire administration; Other: Ancillary studies
- Healing touch therapy following daily radiation (Experimental): All Healing Touch sessions will be given individually, and will be provided by trained nurses or research assistants. Patients receiving Healing Touch will receive a series of standardized therapeutic techniques designed to promote optimal flow of energy throughout the body.
  Interventions: Behavioral: Therapeutic touch; Other: Questionnaire administration; Other: Ancillary studies
- No intervention (Active Comparator): The no intervention group will receive no special intervention other than standard medical care, which includes the regular medical care given by the patient's physician and health care professionals.
  Interventions: Other: Questionnaire administration; Other: Ancillary studies

INTERVENTIONS:
Behavioral: Relaxation training — Muscle relaxation training
  Other Names: Relaxation
  Arms: Relaxation training following daily radiation
Behavioral: Therapeutic touch — Healing Touch (HT) therapy
  Other Names: Healing touch
  Arms: Healing touch therapy following daily radiation
Other: Questionnaire administration
Other: Ancillary studies — Subjects in all groups will give 4 blood samples during the study
  Other Names: Blood draw

SUMMARY:
The proposed project will examine the effects of a healing touch intervention in women receiving chemotherapy and radiation for advanced cervical cancer.

DETAILED DESCRIPTION:
Patients receiving chemoradiation for cervical cancer are at risk for distress, chemoradiation-related side effects, and immunosuppression. This prospective randomized clinical trial proposes to examine the effects of a complementary therapy, Healing Touch (HT), versus relaxation training (RT) and usual care (UC) for (1) supporting cellular immunity, (2) improving mood and quality of life (QOL), and (3) reducing treatment-associated toxicities and treatment delay in cervical cancer patients receiving chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage I-IVa cervical cancer pursuing concurrent chemotherapy and radiation therapy.

Exclusion Criteria:

* Greater than Stage IVa cervical cancer
* Metastatic or recurrent cervical cancer
* Patients receiving only chemotherapy or only radiation therapy
* History of cancer of any site
* History of a transplant
* Diagnosed with any immunosupressive disorder (HIV, AIDS).

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-06-04 (Actual); Primary Completion 2008-03-15 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in natural killer cell cytotoxicity (NKCC) | 6 weeks
  Compare change in natural killer cell cytotoxicity of participants receiving HT during radiation and chemotherapy to participants receiving relaxation training or usual care during radiation and chemotherapy treatment collected via blood draw.
  Fresh peripheral blood mononuclear cells tested for cytolytic activity against the NK-sensitive K562 cells and the NK-resistant LAK-sensitive ZKBL cells in a standard 4-h 51Chromium- release assay.
Number of chemoradiation-related toxicities | 6 weeks
  Compare number of reported side effects of participants receiving HT during radiation and chemotherapy treatment to participants receiving relaxation training or usual care as measured by the Common Toxicity Criteria Manual Version 2.0
Number of days of treatment delay due to chemoradiation-related toxicities | 6 weeks
  Compare number of days in treatment delay due to chemoradiation-related toxicity for participants receiving HT during radiation and chemotherapy treatment to participants receiving relaxation training or usual care
Change in participant reports of depression | 6 weeks
  Compare changes in depression scores of participants receiving HT to participants receiving relaxation training or usual care during radiation and chemotherapy as measured by the Center for Epidemiologic Studies Depression Scale (CES-D) in which higher scores indicate worse depression (range 0-60)

SECONDARY OUTCOMES:
Change in participant reports of anxiety | 6 weeks
  Compare changes in reported anxiety of participants receiving HT during radiation and chemotherapy to participants receiving relaxation training or usual care during radiation and chemotherapy treatment as measured by the Profile of Mood States- Anxiety Subscale (POMS-SF) (range 0-28)
Change in white blood cell counts | 6 weeks
  Compare change in white blood cell counts of participants receiving HT during radiation and chemotherapy vs. patients receiving relaxation training or usual care during this time
  hemotherapy to participants receiving relaxation training or usual care during radiation and chemotherapy treatment collected via blood draw.
Change in red blood cell counts | 6 weeks
  Compare change in red blood cell counts of participants receiving HT during radiation and chemotherapy to participants receiving relaxation training or usual care during radiation and chemotherapy treatment collected via blood draw.
Change in participant reports of quality of life | 6 weeks
  Compare change in reported quality of life of participants receiving HT during radiation and chemotherapy to participants receiving relaxation training or usual care during radiation and chemotherapy treatment as measured by the Functional assessment of Cancer therapies (FACT). Higher scores indicate better quality of life. Range= (0-136).
Change in participant reports of fatigue | 6 weeks
  Compare reported fatigue of participants receiving HT during radiation and chemotherapy to participants receiving relaxation training or usual care during radiation and chemotherapy treatment as measured by the Fatigue Severity Inventory (FSI). Mean fatigue intensity (range 0-10) with higher scores indicating more fatigue, and fatigue duration in days last week experiencing fatigue (0-7 days) with greater number of days indicating greater fatigue duration.
Change in metabolomic measures | 6 weeks
  Compare metabolic profile of participants receiving HT during radiation and chemotherapy treatment to participants receiving relaxation training or usual care. Samples were assayed using Ultrahigh Performance Liquid Chromatography-Tandem Mass Spectroscopy (UPLC-MS/MS). The metabolomic profiling analysis measures the quantity of specific compounds in the plasma vs. a platform of 844 known metabolites in a commercial platform powered by Metabolon, Inc. For any specific metabolite, higher levels indicates greater presence of the metabolite.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Lutgendorf, PhD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lutgendorf SK, Mullen-Houser E, Russell D, Degeest K, Jacobson G, Hart L, Bender D, Anderson B, Buekers TE, Goodheart MJ, Antoni MH, Sood AK, Lubaroff DM. Preservation of immune function in cervical cancer patients during chemoradiation using a novel integrative approach. Brain Behav Immun. 2010 Nov;24(8):1231-40. doi: 10.1016/j.bbi.2010.06.014. Epub 2010 Jun 30. PMID 20600809
- [Background] Hart LK, Freel MI, Haylock PJ, Lutgendorf SK. The use of healing touch in integrative oncology. Clin J Oncol Nurs. 2011 Oct;15(5):519-25. doi: 10.1188/11.CJON.519-525. PMID 21951738